CLINICAL TRIAL: NCT01850316
Title: A Phase II Study for the Treatment of Unresectable or Medically Inoperable Hepatocellular Carcinoma Using Stereotactic Body Radiotherapy (SBRT) in British Columbia
Brief Title: Hepatocellular Carcinoma Using Stereotactic Body Radiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H13-00481
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stereotactic Ablative Radiotherapy (Experimental): Preferred target coverage of 40 Gy: coverage and total dose determined by irradiated liver volume NTCP (normal tissue complication probability) nomogram and OAR dose limits
  Interventions: Radiation: Stereotactic Ablative Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiotherapy — Preferred target coverage of 40 Gy: coverage and total dose determined by irradiated liver volume NTCP (normal tissue complication probability) nomogram and OAR dose limits

SUMMARY:
Respiratory-gated, volumetric-modulated arc therapy will be used for the clinical development of high dose rate Stereotactic Body Radiotherapy (SBRT) in inoperable hepatocellular carcinoma (HCC). These treatments should enhance local control, progression-free survival and potentially overall survival in HCC patients. The investigators will also examine the mechanism of tumour and microenvironmental response to high dose radiation, and search for potential biomarkers to optimize and individualize therapy. Pre-treatment and follow-up PET/CT imaging with 11C-choline, 18F-fluorodeoxyglucose (FDG) and CT perfusion will examine in-vivo changes in proliferation, glycolysis, and the tumour vasculature, respectively, and blood samples will look for immunologic biomarkers of tumour response.

DETAILED DESCRIPTION:
Radiotherapy is not considered standard of care practice for patients for inoperable hepatocellular carcinoma despite the tumour's inherent radiosensitivity. The major challenge has been improving radiation delivery without exceeding dose limits of the surrounding normal liver. Recent technological advances with tumour localization and targeting, imaging, treatment planning and delivery have allowed for safe delivery of radiation with tumorcidal effect and minimal treatment-related toxicity.

This study has three specific aims:

1. To develop, validate, and quality test HDR Stereotactic Body Radiotherapy (SBRT) Gated RapidArc technique for application in human liver tumours. And furthermore, to test whether HDR SBRT Gated RapidArc can be efficiently and safely delivered to a very large patient population previously ineligible for any therapy (HCC patients with tumours >5cm).

3. To determine if 11C-choline/18F-FDG CT-PET or perfusion CT imaging (that characterize changes in tumour proliferation, glycolysis, and vasculature, respectively) can provide practical non-invasive biomarkers of tumour response, local tumour control, or normal tissue toxicity.

4. To determine if immunologic studies of pre- and post-treatment blood samples can provide biomarkers of tumour response, local and systemic tumour control, or triggers for normal tissue toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Multi-phase CT scan of the liver within 8 weeks of radiation planning demonstrating:

   * Liver tumours must be > 5 cm
   * No more than 5 discrete liver tumours may be present
   * Normal liver > 700 cc
3. FDG-PET scan within 12 weeks prior to radiation planning
4. Patients must have HCC diagnosed by either: i) pathological confirmation, or ii) intrahepatic vascular enhancement of the lesion demonstrated by at least two imaging modalities, or iii) intrahepatic vascular enhancement of the lesion demonstrated by one imaging modality if AFP > 200 in the setting of liver cirrhosis or chronic hepatitis B without cirrhosis (EASL consensus guidelines)
5. Liver HCC must be deemed unresectable as determined by an experienced liver surgeon, or the patient must be medically inoperable or refuse surgery, and extra-hepatic metastases must not be present (Patients with potential resectable tumours who are deemed unresectable based on medical inoperability or simultaneous extra-hepatic metastases will be eligible to receive SBRT).
6. Patients must be discussed in a multidisciplinary setting where opinions regarding radiofrequency ablation, various embolotherapies, and targeted biologics are considered, but not eligible for. Patients must have recovered from the effects of previous therapies before SBRT.
7. Eastern Clinical Oncology Group performance status 0,1 or 2 or a Karnofsky performance status of ≥ 60
8. Adequate organ function as assessed by the following blood work:

   * Hemoglobin ≥ 90 g/L
   * Absolute neutrophil count ≥ 1.0 bil/L
   * Platelets ≥ 50 bil/L
   * AST and ALT not to exceed 2x upper limit of normal
9. Child-Turcotte-Pugh assessment (within 8 weeks of treatment date):

   * Bilirubin ≤ 3 mg/dL (< 50 µmol/L)
   * Albumin above 28 g/L
   * INR < 1.7 and/or correctable with vitamin K (unless on anticoagulation therapy)
   * No ascites or encephalopathy
   * Child-Turcotte-Pugh score must be ≤ 7 (see Table 1 in Section 2.1)
10. BCLC Stage B or C (portal venous invasion or liver hilum nodal disease only)
11. No extra-hepatic disease and life expectancy > 6 months
12. No chemotherapy concurrent with radiotherapy
13. Previous treatment(s) with radiofrequency ablation, surgery, TACE, Y90, percutaneous ethanol injection, or chemotherapy are not exclusion criteria provided that recurrence has been documented.
14. Patient signs a study-specific informed consent form. If the patient's mental status precludes this, written informed consent may be given by the patient's legal representative. A translator will be provided if the patient has a language barrier.
15. Treatment plans meet acceptable dose constraints and Liver Veff is ≤ 0.55

Exclusion Criteria:

1. Patients with active hepatitis, encephalopathy, or ascites related to liver failure
2. Female patients who are pregnant (verify with blood test if patient is pre-menopausal). Pre-menopausal patients may also not become pregnant during participation in this study.
3. Prior external beam radiation to the upper abdomen
4. Patients with distant metastases or extrahepatic nodal progression (patients with portal venous thrombosis and liver hilum nodal involvement remain eligible)
5. Patients who have < 700 cc of normal liver.
6. Child-Turcotte-Pugh scores > 7
7. BCLC Stage A, C (N1 and/or M1), D
8. Prior gastric, duodenal, or variceal bleed within the past 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-07; Primary Completion 2018-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
One year local progression-free rate | Approximately 1 year

SECONDARY OUTCOMES:
Progression-free survival | To be reviewed in approximately 8 years; upon study completion
Overall Survival | To be reviewed in approximately 8 years; upon study completion
Treatment related toxicity | To be reviewed in approximately 8 years; upon study completion
Quality of Life | To be reviewed in approximately 8 years; upon study completion
Cytokine response to radiation and association with complications | To be reviewed in approximately 8 years; upon study completion
Functional imaging with 11C-choline/18F-FDG CT-PET and perfusion CT to that characterize treatment-related effects | To be reviewed in approximately 8 years; upon study completion

CONTACTS AND LOCATIONS:
Overall Officials: Roy Ma, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Agency, Vancouver, British Columbia, Canada